CLINICAL TRIAL: NCT07347847
Title: Impact on Mortality of Hospitalisation of a Patient in a Hospital Bed That Does Not Correspond to His Needs After a Visit to the Emergency Department
Acronym: RIGHT BED
Status: Not yet recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC25_30013
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Emergency Department Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
The aim of this study is to assess the impact of hospitalisation outside the referral requested by the emergency doctor on the mortality of patients admitted to emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at an emergency department participating in the study,
* Requiring hospitalisation

Exclusion Criteria:

* Patients hospitalised in short-stay units with secondary outpatient care,
* Adults subject to legal protection (legal guardianship, curatorship, trusteeship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - People Presenting at an emergency department
Sampling Method: Non-Probability Sample
Enrollment: 2766 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Death rate | 30 days

SECONDARY OUTCOMES:
Duration of hospitalization | 30 days
length of stay in the emergency department | 30 days
Rate of Adverse events | 30 days
  Adverse events occuring during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: François Saget, Study Chair — francois.saget@chu-rennes.fr
Locations (7):
- France (7):
  - CHU Angers, Angers
  - CH Le Mans, Le Mans
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours